CLINICAL TRIAL: NCT00004415
Title: Study of Combined Intercostal and Diaphragm Pacing for Artificial Respiration in Quadriplegic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13307; CWRU-09169-M-91; CWRU-FDR000403
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2002-09

CONDITIONS: Quadriplegia
Keywords: environmental/toxic disorders; neurologic and psychiatric disorders; rare disease; spinal cord injury
MeSH Terms: conditions — Quadriplegia; Neurologic Manifestations; Mental Disorders; Rare Diseases; Spinal Cord Injuries

INTERVENTIONS:
Device: Medlink spinal cord electrode

SUMMARY:
OBJECTIVES: I. Determine whether combined intercostal muscle and diaphragm pacing can maintain full-time ventilatory support in patients with ventilatory dependent quadriplegia who are not candidates for phrenic nerve pacing alone.

II. Evaluate the efficacy of the Medlink device to produce synchronous intercostal and diagram activation in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients have a Medlink spinal cord electrode surgically implanted and attached to a radiofrequency receiver implanted subcutaneously over the anterior chest wall.

If substantial inspired volumes can be generated by intercostal pacing, a phrenic nerve cuff electrode and radiofrequency receiver are implanted, and patients undergo combined intercostal muscle and diaphragm pacing.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Ventilator dependent quadriplegics who are not candidates for phrenic nerve pacing alone

Must have bilateral partial or unilateral phrenic nerve function

Must have been on ventilator support for at least 6 months and unweanable

--Patient Characteristics--

Cardiovascular: No active cardiovascular disease

Pulmonary: No active lung disease

Other: No active brain disease Stable condition

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5
Dates: Start 1991-05; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F. DiMarco, Study Chair — Case Western Reserve University